CLINICAL TRIAL: NCT03401138
Title: Preoperative Hemodynamic Monitoring and Resuscitation in Hip Fractures: a Prospective Observational Study
Brief Title: Hemodynamic Monitoring and Resuscitation in Hip Fractures
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Agerskov, MD, Reseach Fellow, Hvidovre University Hospital
Other Study IDs: H- 17037633
Record Dates: First submitted 2018-01-03; First posted 2018-01-17 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Fracture of Hip
Keywords: Peripheral perfusion; Blood Volume; Tissue Prefusion; Near-infrared spectroscopy; Hemodynamic monitoring; Hemodynamic optimization; Preoperative resuscitation
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Preoperative Stroke Volume(SV)-guided fluid optimization — Preoperative SV-guided hemodynamic optimization will be commenced with patients receiving 250ml fluid challenges over five minutes aiming to maximize SV. Maximal SV is defined as absence of a sustained rise in SV by at least 10% in response to a fluid challenge.
  PPI will be obtained from the Masimo Radical 7 (Masimo, Irvine, CA, USA) and NIRS from Invos 5100C (Medtronic, Minneapolis, MN, USA).
  BV measurements will use pulse dye densitometry (PDD) with Indocyanine Green (ICG). We will use the Dye Densitogram 3300 analyser Nihon Kohden (Tokyo, Japan) for registration of the spectrophotometrical absorption of ICG and calculation of BV.
  Other Names: Blood volume measurement; Monitoring of Peripheral Perfusion Index (PPI); Monitoring of Near-infrared Spectroscopy (NIRS)

SUMMARY:
Background: Fracture of the hip is a potentially fatal event in an elderly, frail, highly comorbid patient group suffering from dehydration and hypovolemia, and it carries a risk that equals major trauma in young patients in regard of physiological insult and severity, yet no preoperative resuscitation and transfusion strategy is available. An important goal of hemodynamic monitoring and resuscitation is early detection of insufficient tissue perfusion and oxygenation. The peripheral perfusion index reflects changes in peripheral perfusion and blood volume and a decreased peripheral perfusion index predicts surgical complications and morbidity in acute surgical and septic shock patients. The research group hypothesize that elderly frail patients with a fracture of the hip suffer from hypovolemia and peripheral hypoperfusion of varying degrees and accordingly respond to controlled fluid resuscitation and that the non-invasive peripheral perfusion index will serve as an early predictor of a deteriorated circulation in reflection of stroke volume.

Methods: The main objective of this prospective observational study is to assess to what extend patients with fracture of the hip suffer from hypovolemia and respond to a fluid challenge. The secondary objectives are to evaluate correlation between the minimally-invasive measurements of stroke volume and blood volume and the non-invasive measurement of peripheral perfusion index and near-infrared spectroscopy, as well as prevalence of postoperative complications and mortality. Fifty consecutive patients over the age of 65 years, presenting with a hip fracture, treated in a multimodal fast-track regimen, will be included when written informed consent is available. All patients will receive epidural analgesia and preoperative stroke volume-guided hemodynamic optimization. Blood volume measurements are performed and all patients are monitored with peripheral perfusion index and near-infrared spectroscopy.

Discussion: This is likely the first study to address clinically applicable hemodynamic monitoring and resuscitation in patients with fracture of the hip where adequate resuscitation is easily missed. The study group aim to evaluate the feasibility of preoperative stroke volume-guided hemodynamic optimization in the context of minimally- and non-invasive monitoring of peripheral perfusion and blood volume measurements.

ELIGIBILITY:
Inclusion Criteria:

* Primary acute hip fracture
* Age grater than 65 years
* Written informed consent

Exclusion Criteria:

- Contraindications to epidural analgesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients presenting a primary acute HF within the study period will be screened for participation by the attending anesthesiologist at the post-anesthesia care unit. The study manager will verify the inclusion and exclusion criteria and inform patients (verbally and in writing) and confirm their agreement to participate by asking them to sign the informed consent document. Assessment of electronic patient records, monitoring and resuscitation treatment and recording of data will be by the study manager.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients presenting with preoperative hypovolemia/reduced BV before and after epidural anesthesia | Preoperatively
Proportion of patients with low/very low PPI (PII<1.4 and < 0.5) before and after epidural anesthesia | Preoperatively
Proportion of patients who respond to a 250 ml fluid challenge with sustained rise in SV by at least 10% | Preoperatively

SECONDARY OUTCOMES:
Correlation between SV, PII and NIRS at normo- and hypovolemia states | Preoperatively
Correlation between PPI and standard microcirculatory variables including lactate, capillary refill time (CRT), and central vs. peripheral temperature | Preoperatively
Correlation between non-invasive Hemoglobin (Hb), BV and arterial Hb | Preoperatively
Proportion of mortality in patients responding to the fluid challenge vs. patients not responding | At 30 days and 1 year
Proportion of postoperative complications in patients responding to the fluid challenge vs. patients not responding | At 30 days and 1 year
Proportion of mortality in patients with high vs. low PPI and NIRS, including impact of BV | At 30 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Bang Foss, Clinical Professor, Study Director — Department of Anesthesia, Hvidovre Hospital; Jakob Højlund, MD, Senior Hospital Physiscian, Study Chair — Department of Anesthesia, Hvidovre Hospital; Henrik Sørensen, MD, DMSc, Study Chair — Abdominal Centre, Department of Anesthesia, Rigshospitalet; Niels Secher, Professor, DMSc, Study Chair — Abdominal Centre, Department of Anesthesia, Rigshospitalet; Marianne Agerskov, MD, Research Fellow, Principal Investigator — Department of Anesthesia, Hvidovre Hospital
Locations (1):
- Department af Anesthesia, Hvidovre Hospital, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agerskov M, Sorensen H, Hojlund J, Secher NH, Foss NB. Pre-operative haemodynamic monitoring and resuscitation in hip fracture patients: Protocol for a prospective observational study. Acta Anaesthesiol Scand. 2018 Oct;62(9):1314-1320. doi: 10.1111/aas.13163. Epub 2018 May 30. PMID 29851062